CLINICAL TRIAL: NCT07070674
Title: A Phase Ib Clinical Trial to Investigate the Safety, Tolerability, Preliminary Efficacy, and Pharmacokinetic Profile of AC-003 Capsules in Patients With Acute GraftVersus-Host Disease (aGVHD)
Brief Title: A Phase Ib Clinical Study of AC-003 Capsules in Subjects With aGVHD.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Accro Bioscience (Suzhou) Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AC-003 -CN-PhIb
Record Dates: First submitted 2025-06-30; First posted 2025-07-17 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Acute Graft-versus-Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AC-003 cohort 1 (Experimental): Specified dose of AC-003 will be administered orally twice daily (BID) for 28 days.
  Interventions: Drug: AC-003
- AC-003 cohort 2 (Experimental): Specified dose of AC-003 will be administered orally once daily (QD) for 28 days.
  Interventions: Drug: AC-003
- AC-003 cohort 3 (Experimental): Specified dose of AC-003 will be administered orally twice daily (BID) for 28 days.
  Interventions: Drug: AC-003
- AC-003 cohort 4 (Experimental): Specified dose of AC-003 will be administered orally twice daily (BID) for 28 days.
  Interventions: Drug: AC-003

INTERVENTIONS:
Drug: AC-003 — AC-003 capsules will be administered orally.

SUMMARY:
The study was an open-label, single-arm, dose-escalation, Phase Ib, multi-center study to investigate safety, pharmacokinetics, pharmacodynamics and preliminary efficacy of AC-003 in patients with grade II-IV SR-aGVHD.

DETAILED DESCRIPTION:
The study will enroll approximately 24 subjects in 2 parts:

Part A is a dose-escalation stage to investigate 4 cohorts of AC-003 in adult patients with grade II-IV SR-aGVHD who have undergone allogeneic hematopoietic stem cell transplantation.

The dose escalation will start with cohort 1, in which patients will receive specified dose of AC-003 capsules orally for 28 days and escalate to cohort 2, 3 and 4 sequentially when the previous cohort is deemed to be safe by Safety Review Committee (SRC). Safety follow-up will occur on Day 35. Decision of recommended dose will be made depend on the safety, PK and PD assessments across cohorts.

Part B is a dose-expansion stage to investigate the preliminary efficacy of recommended dose. Patient will receive recommended dose of AC-003 capsules orally for 28 days. Safety follow-up will occur on Day 35.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age ≥ 18 years.
2. Patients who have undergone allogeneic hematopoietic stem cell transplantation (HSCT) from any donor source (including matched unrelated donor, haplo-identical).
3. Diagnosis of grade II-IV aGVHD as per MAGIC criteria within 100 days after HSCT.
4. Diagnosis of steroid-refractory or steroid-dependent aGVHD in at least one of the following criteria:

   1. Progressive Disease, defined as any target organ worsening, after 3 days of initial treatment with methylprednisolone 1~2 mg/kg/day (or equivalent corticosteroid)
   2. Not partial response after 7 days of initial treatment with methylprednisolone 1~2 mg/kg/day (or equivalent corticosteroid)
   3. Not complete response after 14 days of initial treatment with methylprednisolone 1~2 mg/kg/day (or equivalent corticosteroid)
   4. Relapse of aGVHD when corticosteroid tapering.

Exclusion Criteria:

1. Evidence of aGVHD relapsed.
2. Evidence of chronic GVHD or overlap syndrome
3. Receipt of more than one allogeneic HSCT
4. Receipt of more than one systemic treatment for aGVHD in addition to corticosteroid
5. Any corticosteroid therapy for indications other than aGvHD at doses >= 1 mg/kg/day methylprednisolone (or equivalent corticosteroid) within 7 days prior to enrolment
6. Severe organ dysfunction unrelated to aGVHD
7. Uncontrolled active infection (i.e., bacterial, fungal, or viral)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events | Up to Day 35
  An Adverse Event (AE) is defined as any new untoward medical condition or worsening of a pre-existing medical condition following or during exposure to an investigation product, whether or not considered causally related to the product.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Day 14 and Day 28
  ORR is the percentage of patients with complete response (CR) or partial response (PR) as determined by investigator.
  CR is defined as all target organs evaluated as Mount Sinai Acute GVHD International Consortium (MAGIC) Stage 0 [Skin - no active GVHD rash; Liver - bilirubin <2 mg/dL; Upper gastrointestinal (GI) tract - no intermittent nausea, vomiting/anorexia; Lower GI tract - stool output: < 500 mL/day or <3 episodes/day (adults)].
  PR is defined as improvement in one or more target organs (skin, liver, upper GI tract, lower GI tract) involved with aGVHD symptoms without worsening in others.
Complete Response Rate | Day 14 and Day 28
  Complete Response Rate is the percentage of patients with complete response (CR).
  CR is defined as all target organs evaluated as Mount Sinai Acute GVHD International Consortium (MAGIC) Stage 0 [Skin - no active GVHD rash; Liver - bilirubin <2 mg/dL; Upper gastrointestinal (GI) tract - no intermittent nausea, vomiting/anorexia; Lower GI tract - stool output: < 500 mL/day or <3 episodes/day (adults)].

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Hospital of Chinese Academy of Medical Sciences (Institute of Hematology, Chinese Academy of Medical Sciences), Tianjin, Tianjin Municipality, China